CLINICAL TRIAL: NCT01627470
Title: Evaluation of a Continuous Non-invasive Arterial Pressure Device in Comparison With Invasive Pressure Measurement During Out-of-hospital Emergency
Brief Title: Comparison of Continuous Non-invasive Pressure Device Versus Invasive Pressure Measurement During Prehospital Emergency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Robert Hanss (Other)
Responsible Party: Sponsor-Investigator, Robert Hanss, PD Dr. med., University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Other Study IDs: CNAP-ITW
Record Dates: First submitted 2011-11-02; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Blood Pressure
Keywords: non-invasive arterial pressure; emergency; intensive care
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Emergency Patients with applied arterial blood pressure measurement
  Interventions: Device: CNAP-Monitor

INTERVENTIONS:
Device: CNAP-Monitor — Continuous non-invasive arterial blood pressure recording
  Other Names: CNAP; Continuous non-invasive arterial blood pressure recording

SUMMARY:
The aim of the study is to evaluate the accuracy of continuous non-invasive AP monitoring (CNAP) compared to simultaneous IBP measurement in intensive care patients undergoing a transport in the ambulance car.

Since CNAP finger blood pressure is calibrated to NBP level, a systematic bias between IBP and CNAP as described by a recent FDA meta analysis [ ] is expected. The most important factor of CNAP system performance is its ability to accurately track blood pressure changes. Thus, the purpose of this investigation is to show that the bias between CNAP and IBP falls within the expected range and that blood pressure alterations are detected instantaneously.

The endpoints of the study are:

* The agreement of systolic, diastolic and mean CNAP and IBP readings determined on a beat-to-beat basis during:
* Takeover of the patient on the intensive care unit,
* Transport of the patient from the intensive care unit to the ambulance car
* Transport of the patient in the ambulance car
* The agreement of systolic, diastolic and mean CNAP and IBP blood pres-sure changes determined on a beat-to-beat basis during:
* Takeover of the patient on the intensive care unit,
* Transport of the patient from the intensive care unit to the ambulance car
* Transport of the patient in the ambulance car

The beat-to-beat readings of CNAP and IBP will be automatically recorded electronically on a memory card in the transport monitor. CNAP data will additionally be recorded directly on the CNAP Monitor with a memory stick. Safety will be assessed by clinical observations as well as adverse events (AE) recording.

DETAILED DESCRIPTION:
Arterial pressure (AP) is one of the most important physiological variables. Particularly in emergency medicine, AP needs to be monitored repeatedly or even better, continuously. This is usually done using an oscillometric pressure device (NIBP). A number of studies emphasise the importance of continuous AP monitoring as more than 20% of all hypotensive episodes may be missed by NIBP and another 20% are detected with delay. Prolonged hypotension precedes 56% of perioperative cardiac arrests and is associated with a significant increase of the 1-year mortality rate, indicating that NBP monitoring especially in patients with cardiovascular diseases might be insufficient independent from the clinical setting. Recently, a monitor for continuous non-invasive AP monitoring (CNAP™ Monitor 500) was introduced. It was shown that during procedures with high risk of hypotension NIBP missed significant more hypotensive episodes than CNAP. At the moment we have no evidence of the performance of CNAP in the preclinical emergency medicine. The evaluation against the gold standard of invasive pressure measurement in this study will help us to evaluate the performance of CNAP in the preclinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and capable of giving informed consent or with legal agents willing of giving informed consent
* Patients undergoing a transport from the intensive care unit to another institution with the ambulance car
* Patients where the IBP cannula was already placed on the intensive care unit
* Patients where IBP cannula, and CNAP upper arm cuff can be placed on the same arm, and CNAP finger cuff can be placed on the contra-lateral arm
* Intact perfusion of both arm evidenced by a negative Allen's test
* Age 18 years and above
* ASA I-IV
* Weight >= 40 and <= 180 kg, BMI < 35

Exclusion Criteria:

* Patients with history of neurological, neuromuscular seizure
* Patients where IBP cannula cannot be placed in the radial artery
* Patients with vascular implants at the sites of non-invasive blood pressure measurement (fingers and upper arm)
* Patients with history of arrhythmias
* Edematous patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU Patients with established arterial pressure measurement
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
agreement with invasive blood pressure | 1 year
  beat-to-beat readings of CNAP and IBP

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hanss, PD Dr., Study Chair — UKSH-Campus Kiel
Locations (1):
- University Hospital Schleswig-Holstein - Campus Kiel, Kiel, Germany